CLINICAL TRIAL: NCT06132360
Title: A Phase 1, Randomized, Single-blinded, Placebo-controlled, Single-ascending-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects in Adult Subjects With Elevated LDL-C
Brief Title: the Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects in Adult Subjects With Elevated LDL-C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Rona Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RN0191-102
Record Dates: First submitted 2023-11-06; First posted 2023-11-15 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2023-11

CONDITIONS: To Reduce the LDL-C Level in Hypercholesteremia Patients

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cohort 1 (Experimental): or placebo
  Interventions: Drug: RN0191
- Cohort 2 (Experimental): or placebo
  Interventions: Drug: RN0191
- Cohort 3 (Experimental): or placebo
  Interventions: Drug: RN0191
- Cohort 4 (Experimental): or placebo
  Interventions: Drug: RN0191

INTERVENTIONS:
Drug: RN0191 — This is a randomized, placebo-controlled, single ascending-dose (SAD) study of RN0191 administered SC to adult subjects with elevated LDL-C. Subjects who have signed an Ethics Committee (EC)-approved informed consent form (ICF) and have met all the protocol eligibility criteria during screening may be enrolled into the study.

SUMMARY:
This is a randomized, placebo-controlled, single ascending-dose (SAD) study of administered SC to adult subjects with elevated LDL-C. Subjects who have signed an Ethics Committee (EC)-approved informed consent form (ICF) and have met all the protocol eligibility criteria during screening may be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, aged 18 to 60 years, inclusive
2. Body mass index between 18 and 32 kg/m2, inclusive, with body weight > 45 kg for females and >50 kg for males
3. Serum LDL-C ≥100 mg/dL (2.6 mmol/L) at screening and Day -1
4. Fasting triglycerides < 400 mg/dL (<4.52 mmol/L) at screening and Day -1

Exclusion Criteria:

1. Known underlying disease or medical condition that may have a potential impact on general safety assessment, lipid metabolism, or glucose metabolism, or surgical condition (including, but not limited to, bariatric surgery) that, in the opinion of the investigator, may interfere with the interpretation of the results of the clinical study
2. Received any medication including, but not limited to, statins, ezetimibe, or lipid-altering nutrients within 30 days prior to screening, or PCSK9 antibody within 90 days prior to screening, or any LDL-C-lowering siRNA therapy within 12 months prior to screening
3. History of multiple drug allergies or allergic reactions to oligonucleotides or N-acetylglucosamine (GalNAc)
4. Subjects with alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 1.5 times the upper limit of normal (ULN) at the time of screening (one repeat of the screening assay is permitted) with clinically significant ALT and/or AST > ULN and ≤ 1.5 times the ULN as determined by the investigator
5. Any medical condition that, in the opinion of the Investigator, makes the subject unsuitable for enrollment or may interfere with the subject's participation in or completion of the study. This includes, but is not limited to: history or presence of cardiovascular disease (including peripheral arterial and cerebrovascular disease); diabetes mellitus (except for diabetes mellitus of pregnancy in remission); cerebrovascular accidents; and abnormal thyroid function.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of RN0191 administered as escalating single subcutaneous (SC) doses in adult subjects with elevated low-density lipoprotein-cholesterol (LDL-C) | For each subject in the study, the duration of the study clinic visits is approximately 18 weeks from screening to Day 85 EOS examination.
  This is a randomized, placebo-controlled, single ascending-dose (SAD) study of RN0191 administered SC to adult subjects with elevated LDL-C. Subjects who have signed an Ethics Committee (EC)-approved informed consent form (ICF) and have met all the protocol eligibility criteria during screening may be enrolled into the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China